CLINICAL TRIAL: NCT07349420
Title: CLEC10A-Targeted M2 Macrophage Repolarization With EF-M2 (Immutalon) in Patients With Moderate-to-Severe Rheumatoid Arthritis: An Open-Label, Multicenter, First-in-Human Phase I/IIa Multiple Ascending Dose Study
Brief Title: EF-M2 (Immutalon) Multiple Ascending Dose Study in Moderate-to-Severe Rheumatoid Arthritis
Acronym: MACRA-FIH-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Activator MAF, LLC (Unknown); Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SW032
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: EF-M2; Immutalon; Multiple Ascending Dose; Macrophage Repolarization
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Open-label, multiple ascending dose study with sequential cohort dose escalation. Participants receive EF-M2 (Immutalon) by subcutaneous injection for 4 weeks (twice weekly in Cohorts 1-4). Optional expanded pharmacodynamic cohorts may evaluate increased dosing frequency (three times weekly). Sentinel dosing is used at the start of each new cohort, and dose escalation proceeds after DSMB review of safety and pharmacodynamic data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1: EF-M2 1 mcg SC Twice Weekly (Experimental): Participants receive EF-M2 (Immutalon) 1 mcg by subcutaneous injection twice weekly for 4 weeks (8 injections total).
  Interventions: Drug: EF-M2
- Cohort 2: EF-M2 3 mcg SC Twice Weekly (Experimental): Participants receive EF-M2 (Immutalon) 5 mcg by subcutaneous injection twice weekly for 4 weeks (8 injections total).
  Interventions: Drug: EF-M2
- Cohort 4: EF-M2 7 mcg SC Twice Weekly (Experimental): Participants receive EF-M2 (Immutalon) 7 mcg by subcutaneous injection twice weekly for 4 weeks (8 injections total).
  Interventions: Drug: EF-M2
- Cohort 5: EF-M2 3 mcg SC Three Times Weekly (Experimental): Participants receive EF-M2 (Immutalon) 3 mcg by subcutaneous injection three times weekly for 4 weeks (12 injections total). Optional expanded pharmacodynamic cohort.
  Interventions: Drug: EF-M2
- Cohort 6: EF-M2 5 mcg SC Three Times Weekly (Experimental): Participants receive EF-M2 (Immutalon) 5 mcg by subcutaneous injection three times weekly for 4 weeks (12 injections total). Optional expanded pharmacodynamic cohort.
  Interventions: Drug: EF-M2
- Cohort 3: EF-M2 5 mcg SC Twice Weekly (Experimental): Participants receive EF-M2 (Immutalon) 5 mcg by subcutaneous injection twice weekly for 4 weeks (8 injections total).
  Interventions: Drug: EF-M2

INTERVENTIONS:
Drug: EF-M2 — EF-M2 (Immutalon) is an investigational product administered as a subcutaneous injection. In this study, participants receive EF-M2 for 4 weeks in sequential multiple ascending dose cohorts: 1, 3, 5, or 7 mcg twice weekly (8 injections total). Optional expanded pharmacodynamic cohorts may receive 3 or 5 mcg three times weekly (12 injections total).

SUMMARY:
This is a first-in-human, open-label, phase I/IIa, multiple ascending dose study of EF-M2 (Immutalon), a macrophage-modulating investigational product intended to shift macrophages toward an anti-inflammatory (M2-like) phenotype via a CLEC10A-mediated mechanism. The study will enroll adults with moderate-to-severe rheumatoid arthritis.

Participants will receive EF-M2 as subcutaneous injections for 4 weeks in sequential dose cohorts (1, 3, 5, or 7 mcg administered twice weekly; optional expanded pharmacodynamic cohorts may receive 3 or 5 mcg three times weekly). The total number of injections will be 8-12 depending on the regimen. Dose escalation is sequential and overseen by an independent data safety monitoring board (DSMB), with sentinel dosing at the start of each new cohort. Participants may be followed off drug for up to 8-12 weeks after treatment, for a total participation time of up to 16 weeks (including screening).

The primary objective is to evaluate safety, tolerability, and immunogenicity. Secondary objectives include assessing pharmacodynamic markers of M2 polarization (e.g., changes in ARG1/iNOS and IL-10/TNF-α ratios and M2-associated cell phenotypes) and exploring associations with clinical activity measures.

DETAILED DESCRIPTION:
This phase I/IIa, open-label, multicenter, multiple ascending dose (MAD) study evaluates EF-M2 (Immutalon) administered subcutaneously to adults with moderate-to-severe rheumatoid arthritis. The trial is designed primarily to characterize safety/tolerability and immunogenicity and to describe pharmacodynamic (PD) evidence of macrophage M2 polarization rather than to demonstrate definitive clinical efficacy.

Participants are enrolled into sequential dose cohorts. Each participant receives EF-M2 for 4 weeks: Cohorts 1-4 receive 1, 3, 5, or 7 mcg twice weekly (8 injections total). If needed, expanded PD cohorts may evaluate 3 mcg or 5 mcg administered three times weekly (12 injections total) to better understand whether increased dosing frequency strengthens the M2 PD signature and where a plateau may begin. Dose escalation is sequential and occurs only after DSMB review of safety and PD data; sentinel dosing is used in each new cohort (the first 2 participants receive initial dosing with an observation period before full cohort enrollment continues).

Key assessments include adverse event monitoring, physical examinations and vital signs at visits, laboratory safety testing at scheduled time points, and immunogenicity testing (anti-drug antibodies, with neutralizing antibodies assessed if antibodies are detected). Pharmacodynamic assessments are based on blood markers measured over time (e.g., soluble cytokines and macrophage/monocyte markers), with PD endpoints including change in ARG1/iNOS and IL-10/TNF-α ratios and changes in M2-associated cell phenotypes.

Study timing includes screening up to 28 days, 4 weeks of treatment, and an off-drug follow-up period of 8-12 weeks (total participation up to 16 weeks). Example follow-up assessments extend through Day 112. The planned sample size is approximately 32 participants (8 per cohort across four dose levels), with up to 48 participants if both expanded PD cohorts are activated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years.
* Diagnosis of rheumatoid arthritis according to the 2010 American College of - Rheumatology and European Alliance of Associations for Rheumatology classification criteria for at least 6 months.
* Moderate-to-severe active disease, defined as:
* Disease Activity Score in 28 joints using C-reactive protein at least 3.2 and not more than 6.0; and
* At least 6 tender joints and at least 6 swollen joints based on the 28-joint count.
* Inadequate response to at least one conventional synthetic disease-modifying antirheumatic drug (for example, methotrexate or leflunomide); and either:
* No prior biologic or targeted synthetic disease-modifying antirheumatic drug therapy; or
* No more than one prior line of biologic or targeted synthetic disease-modifying antirheumatic drug therapy, discontinued at least 12 weeks before screening.
* Stable background therapy:
* Conventional synthetic disease-modifying antirheumatic drug at a stable dose for at least 8 weeks; and
* Glucocorticoids at a dose not exceeding 10 milligrams per day of prednisone (or equivalent) at a stable dose for at least 4 weeks; and
* Nonsteroidal anti-inflammatory drugs and/or analgesics on a stable regimen for at least 2 weeks.
* Willingness and ability to comply with study visits, biospecimen collection, and contraception requirements (for women and men).

Exclusion Criteria:

* Current severe infection; active or latent tuberculosis without completed preventive therapy.
* Chronic hepatitis B, chronic hepatitis C, or human immunodeficiency virus infection with high viral load.
* Active malignancy or history of malignancy within 5 years, except adequately treated carcinoma in situ of the cervix or skin.
* History of severe opportunistic infections.
* Uncontrolled cardiovascular disease (including New York Heart Association class III or IV heart failure, acute coronary syndrome within the past 6 months, or uncontrolled arterial hypertension), decompensated diabetes mellitus, or severe liver or kidney disease.
* Pregnancy, breastfeeding, or planning pregnancy within 6 months.
* Prior treatment with cellular therapies, chimeric antigen receptor T-cell therapy, or profound immunosuppressive therapies with incomplete immune reconstitution.
* Any condition that, in the investigator's opinion, increases the risk of study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-12-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events | From first dose (Day 0) through end of follow-up (Day 112)
  Number and percentage of participants with any treatment-emergent adverse event and with any serious adverse event during the study. Events will be coded and summarized by severity and relationship to study drug; severity will be graded using the Common Terminology Criteria for Adverse Events.
  Range and Units: Count: 0 to total number of participants. Percentage: 0% to 100%.
Incidence of Dose-Limiting Toxicities | From first dose (Day 0) through end of dosing period (Day 28)
  Number and percentage of participants who experience a dose-limiting toxicity during the dose-limiting toxicity evaluation period (pre-defined clinically significant toxicities, including severe toxicities graded using the Common Terminology Criteria for Adverse Events, immune complications, and severe infections as specified by protocol).
  Range and Units: Count: 0 to total number of participants in the cohort. Percentage: 0% to 100%.
Percentage of Participants With Treatment-Emergent Clinically Significant Laboratory Abnormalitie | Baseline (Day 0) and Days 7, 14, 28, 56, 84, and 112
  Treatment-emergent clinically significant laboratory abnormality is defined as a post-baseline abnormality meeting Grade 3 or Grade 4 severity criteria (per CTCAE v5.0, or equivalent protocol-defined grading) in any of the assessed laboratory parameters, including hematology (CBC with differential and platelets), serum chemistry (ALT, AST, alkaline phosphatase, bilirubin, creatinine, urea, electrolytes), inflammatory markers (C-reactive protein, fibrinogen), and immune markers (immunoglobulins and complement).
  A participant will be counted once if they experience ≥1 qualifying abnormality at any post-baseline assessment. Results will be summarized as a percentage of participants.
Proportion of Participants With Anti-Drug Antibodies and Neutralizing Antibodies to EF-M2 | Baseline (Day 0) and Days 28, 56, 84, and 112
  Number and percentage of participants with a positive anti-drug antibody result to EF-M2 in serum. Neutralizing antibodies will be assessed in participants with positive anti-drug antibodies.
  Range and Units: Count: 0 to total number of participants tested. Percentage: 0% to 100%.

SECONDARY OUTCOMES:
Change From Baseline in Arginase 1 to Inducible Nitric Oxide Synthase Ratio | Baseline (Day 0) to Day 28, Day 56, and Day 84
  Change from baseline in the ratio of arginase 1 to inducible nitric oxide synthase measured in enriched peripheral blood monocytes using reverse transcription quantitative polymerase chain reaction. The outcome is expressed as a unitless ratio.
  Range and Units: Unitless ratio; minimum 0; no protocol-defined maximum. Change from baseline can be negative or positive.
Change From Baseline in Plasma Interleukin 10 to Tumor Necrosis Factor Alpha Ratio | (Day 0) to Day 28, Day 56, and Day 84
  Change from baseline in the ratio of plasma interleukin 10 concentration to plasma tumor necrosis factor alpha concentration, measured using multiplex cytokine panels. The outcome is expressed as a unitless ratio.
  Range and Units: Unitless ratio; minimum 0; no protocol-defined maximum. Change from baseline can be negative or positive.
Change From Baseline in Proportion of Monocytes With M2-Associated Phenotype | Baseline (Day 0) to Day 28, Day 56, and Day 84
  hange from baseline in the proportion of peripheral blood monocytes/macrophage-lineage cells with an M2-associated phenotype, defined by expression of mannose receptor C-type 1 (also known as cluster of differentiation 206) and MER proto-oncogene, tyrosine kinase (also known as MerTK), assessed by flow cytometry or mass cytometry within the monocyte population (cluster of differentiation 14 positive, cluster of differentiation 16 plus/minus).
  Range and Units: Percentage: 0% to 100%. Change from baseline can be negative or positive (percentage points).
Pharmacodynamic Differences Between Dose Levels and Dosing Regimens | Baseline (Day 0) to Day 28, Day 56, and Day 84
  Differences between dose levels (1, 3, 5, and 7 micrograms) and dosing regimens (twice weekly versus three times weekly, if expanded cohorts are activated) in change from baseline pharmacodynamic markers of M2 polarization, including (1) arginase 1 to inducible nitric oxide synthase ratio and (2) plasma interleukin 10 to tumor necrosis factor alpha ratio.
  Range and Units: Between-group difference in change from baseline for unitless ratios; no protocol-defined minimum or maximum.
Dose-Pharmacodynamic Relationship for M2 Polarization Markers | Baseline (Day 0) to Day 28, Day 56, and Day 84
  Dose-pharmacodynamic relationship for change from baseline in (1) arginase 1 to inducible nitric oxide synthase ratio and (2) plasma interleukin 10 to tumor necrosis factor alpha ratio, evaluated across dose levels (and dosing frequency if applicable) using nonlinear dose-response modeling (for example, maximum effect models).
  Range and Units: Model-based relationship for unitless ratios; no protocol-defined minimum or maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Technologies, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: No